CLINICAL TRIAL: NCT06093893
Title: A Comparison of Dexmedetomidine, Nicardipine, and Labetalol to Induce Hypotensive Anesthesia and Their Effects on Surgeon Visibility, Blood Loss, Hemodynamic Parameters, Operation Time, and Adverse Events During Orthognathic Surgery
Brief Title: Hypotensive Anesthesia for Orthognathic Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-43663
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypotensive Anesthesia; Orthognathic Surgery
Keywords: Dexmedetomidine; Nicardipine; Labetalol; Surgeon visibility; Blood loss; Hemodynamic parameters; Operation time
MeSH Terms: conditions — Hemorrhage | interventions — Dexmedetomidine; Nicardipine; Labetalol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dexmedetomidine group (Experimental): Participants randomized into this group will be given Dexmedetomidine to lower their blood pressure during jaw surgery.
  Interventions: Drug: Dexmedetomidine
- Nicardipine group (Experimental): Participants randomized into this group will be given Nicardipine to lower their blood pressure during jaw surgery.
  Interventions: Drug: Nicardipine
- Labetalol group (Experimental): Participants randomized into this group will be given Labetalol to lower their blood pressure during jaw surgery.
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg will be administered intravenously over 10 minutes; followed by maintenance infusion of 0.2 to 1 mcg/kg/hour.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Nicardipine — 1 mg will be administered intravenously and increase by 0.5-1 mg if the initial dose is ineffective, to a maximum of 15 mg / hour or
  Other Names: Cardene
  Arms: Nicardipine group
Drug: Labetalol — 20 - 80 mg will be administered intravenously at 10-minute intervals to maximum of 300 mg;
  Other Names: Labetalol hydrochloride injection
  Arms: Labetalol group

SUMMARY:
The overall objective of this double blinded, randomized controlled trial (RCT) is to compare specific outcomes of three medications (Dexmedetomidine, Nicardipine, and Labetalol) which are routinely used to lower blood pressure used during general anesthesia for orthognathic (jaw) surgery. The outcome measures for the study will be surgical field visibility, estimated blood loss, hemodynamic parameters, operation time, and adverse events.

The specific objectives of this study are to compare:

1. Dexmedetomidine, Nicardipine, and Labetalol's effect on the quality of the surgical field. (Primary Outcome)
2. Dexmedetomidine, Nicardipine, and Labetalol's effect on estimated blood loss.
3. Dexmedetomidine, Nicardipine, and Labetalol's effect on hemodynamic parameters including systolic blood pressure, mean arterial pressure, and heart rate.
4. Dexmedetomidine, Nicardipine, and Labetalol's effect on operation time.
5. Dexmedetomidine, Nicardipine, and Labetalol's effect on adverse events.

The investigators will evaluate healthy adult male and female patients who require jaw surgery at Boston Medical Center. The anticipated 90 participants will be randomized into three groups: ) A Labetalol group in which the patients receive hypotensive anesthesia with the aid of labetalol, 2) A Nicardipine group in which the patients receive hypotensive anesthesia with the aid of nicardipine, and 3) A Dexmedetomidine group in which the patients receive hypotensive anesthesia with the aid of dexmedetomidine.

The time it will take for each individual participant ranges from 1-3 months. This time includes the pre-operative visit, the surgical procedure, a 1-week post-operation visit, and then followed for 30 days post-operatively after which the patient's participation in the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing orthognathic surgery [Le Fort I, Surgically Assisted Rapid Palatal Expansion (SARPE), Bilateral Sagittal Split Osteotomy (BSSO), or a combination these surgeries] at Boston Medical Center with Dr. Mehra
* Healthy, American Society of Anesthesiologists (ASA) physical status classification system I or II

Exclusion Criteria:

* Patients on a home beta blocker
* Patients on home calcium channel blocker
* Patients on home alpha 2 agonists
* Patients with an allergy to one or more of the intervention medications
* Does not speak English
* Pregnant patients (this is assessed day of surgery per standard care with a urine pregnancy test)
* Patients who have contraindications to induced hypotensive anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Surgical field visibility | immediately after surgery
  Surgical field visibility will be assessed using the Fromme's scale (0 = no bleeding, virtually bloodless field, 1 = bleeding, so mild it was not even a surgical nuisance, 2= moderate bleeding, a nuisance but without interference with accurate dissection, 3 = moderate bleeding that moderately compromised surgical dissection, 4 = bleeding, heavy but controllable, that significantly interfered with dissection, 5 = massive uncontrollable bleeding). This data will be obtained from the surgeon in the form of an electronic survey, and the mean value will be recorded.

SECONDARY OUTCOMES:
Estimated blood loss | immediately after surgery
  This outcome will be calculated by the volume in suction minus the volume of irrigating fluid.
Mean systolic blood pressure during surgery | throughout surgery every 5 minutes
  This outcome will be automatically recorded in the electronic medical record every 5 minutes during surgery.
Mean arterial pressure | throughout surgery every 5 minutes
  This outcome will be automatically recorded in the electronic medical record every 5 minutes during surgery.
Mean heart rate | throughout surgery every 5 minutes
  This outcome will be automatically recorded in the electronic medical record every 5 minutes during surgery.
Operation time | immediately after surgery
  Operation time will be measured from time of first incision to procedure end, as recorded in electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Pushkar Mehra, DMD, Principal Investigator — Oral and Maxillofacial Surgery Department, Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No